CLINICAL TRIAL: NCT03826381
Title: Prevalence and Metabolic Impact of Non-alcoholic Fatty Liver Disease in Patients With Type 2 Diabetes With Normal Renal Function or Chronic Kidney Disease
Brief Title: NAFLD Among Patients With Type 2 Diabetes and CKD
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, Professor, Rigshospitalet, Denmark
Other Study IDs: NAFLD and CKD - Study 1
Record Dates: First submitted 2018-03-18; First posted 2019-02-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Chronic Kidney Diseases; Type2 Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Renal Insufficiency, Chronic | interventions — Magnetic Resonance Imaging; Continuous Glucose Monitoring; Absorptiometry, Photon; Blood Specimen Collection; Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for both immediately analyses (basic lab data) and later analyses (bile acids,lipidomics and metabolomics) and stored for 10 years whereafter they will be destroyed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study 1: DM2 + normal kidney function: Number of patients: 54
  Patients in this group are diagnosed with Diabetes type 2. Kidney function: eGFR is > 60, absence of clinical proteinuria.
  Inclusion- and exclusion criteria are listed under section "Eligibility". Examinations performed in this group are listed under the section "Groups and Interventions" and the same as in the other group.
  The patients are examined once.
  Interventions: Diagnostic Test: Magnetic resonance (MR) spectroscopy of the liver; Diagnostic Test: Fibroscan; Device: Continuous glucose monitoring (CGM) for four days.; Radiation: Dual Energy X-ray Absorptiometry (DEXA) scan; Biological: Blood samples; Other: Clinical and demographic data
- Study 1: DM2 + CKD stage 3-5: Number of patients: 54
  Patients in this group are all diagnosed with diabetes type 2. Furthermore, the patients have chronic kidney disease stage 3-5 (eGFR <60).
  Inclusion- and exclusion criteria are listed under section "Eligibility". Examinations performed in this group are listed under the section "Groups and Interventions" are the same as in the other group.
  The patients are examined once.
  Interventions: Diagnostic Test: Magnetic resonance (MR) spectroscopy of the liver; Diagnostic Test: Fibroscan; Device: Continuous glucose monitoring (CGM) for four days.; Radiation: Dual Energy X-ray Absorptiometry (DEXA) scan; Biological: Blood samples; Other: Clinical and demographic data

INTERVENTIONS:
Diagnostic Test: Magnetic resonance (MR) spectroscopy of the liver — Magnetic resonance (MR) spectroscopy of the liver. Golden standard for non-invasive determination of NAFLD
Diagnostic Test: Fibroscan — Transient Elastography for Measurement of liver fibrosis.
Device: Continuous glucose monitoring (CGM) for four days. — CGM is attached to the abdominal skin for four days. Afterwards data is converted and analysed in a computer program.
Radiation: Dual Energy X-ray Absorptiometry (DEXA) scan — DEXA-scan of the body composition.
Biological: Blood samples — Immediately analyse of basic lab data. Later analyses for glucagon, amino acids, bile acids, lipidomics and metabolomics.
Other: Clinical and demographic data — Measurements of blood pressure, pulse, height, weight.

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in developed countries affecting approximately 30 % of the general adult population. It represents an important pathogenic factor in the development of type 2-diabetes and is associated with a high risk of cardiovascular disease. Previous studies of patients with chronic kidney disease (CKD) have demonstrated an increased risk for NAFLD and the presence of both CKD and NAFLD is likely to increase the risk for cardiovascular disease.

The present protocol describes a study of the prevalence and etiology of NAFLD among patients with type 2-diabetes with CKD.

The study is a cross-sectional study. Fat accumulation in the liver will be determined by Magnetic resonance (MR) spectroscopy and the prevalence of NAFLD among patients with type 2-diabetes with normal kidney function or CKD stage 3-5 will be investigated. A continuous glucose monitoring (CGM) for four days, Dual Energy X-ray Absorptiometry (DEXA) scanning, fibro scanning of the liver, bile acid analysis, metabolomic and lipidomic analysis will also be performed.

DETAILED DESCRIPTION:
INTRODUCTION

Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in developed countries affecting approximately 30 % of the general adult population. The disease is defined by an increased fat accumulation in the liver cells (>5 %), not caused by excessive alcohol intake (a threshold of 20 g per day for women and 30 g per day for men), autoimmunity, drugs or viral hepatitis. The histological spectrum of NAFLD ranges from simple steatosis to non-alcoholic steatohepatitis (NASH). Simple steatosis defined as steatosis without injury of the hepatocytes in form of ballooning and NASH defined as the presence of hepatic steatosis and inflammation with ballooned hepatocytes with or without fibrosis. The degree of fibrosis is an important prognostic factor and is related to liver related complications and mortality.

Diabetes is the single most important cause of end-stage renal disease (ESRD). Furthermore, more than 25 % of patients with moderate to severe chronic kidney disease (CKD) have pre-diabetic characteristics such as impaired glucose tolerance or impaired fasting glucose. NAFLD represents an important pathogenic factor in the development of type 2-diabetes and is associated with an increased risk of cardiovascular disease, insulin resistance and overweight.

Previous studies of patients with CKD with/without diabetes demonstrated, with less sensitive ultrasonic methods than what we plan to use in the present project, a high prevalence of NAFLD. Furthermore, the presence of both NAFLD and CKD is likely to increase the risk for cardiovascular diseases and mortality, particular among overweight patients. NAFLD is present in both diabetic and nondiabetic patients with ESRD. The co-existence of CKD, NAFLD and gluco-metabolic disturbances, including diabetes, is a research topic with increasing focus on. Co-morbidities in CKD such as impaired insulin sensitivity, diabetes, impaired calcium-phosphate metabolism, hypertension and hypertriglyceridemia constitute risk factors for NAFLD. Unfortunately, several treatments of CKD, including kidney transplantation, have been shown to impair lipid metabolism and increase insulin resistance especially in the liver. Importantly, lifestyle changes and medical treatment modalities have been shown to have only minor impact on reducing the prevalence of these disturbances in patients with CKD.

In patients with NAFLD, either due to metabolic stress (obesity) or toxic substances (immunosuppressive treatment), liver damage and the impact on insulin resistance is reflected in characteristic modifications of metabolites and lipids in liver tissue, as well as in circulating blood, which may help to identify and interpret the pathogenesis of liver damage in the setting of CKD. One recent hypothesis for linking liver damage and CKD involves a change in gut microbiota due to impaired renal function, leading to a leaky gut with damage of the gut-blood barrier. This transfers gut microbiota metabolites to the blood, leading to a pathogen-associated molecular pattern, reflected in changes in lipidomic and metabolomic profile in the blood. Such changes have in other conditions been associated with insulin resistance and have been linked to liver damage leading to NAFLD and later potentially fibrosis.

Very little information about bile acid metabolism in the development of NAFLD in CKD patients with type 2-diabetes is available. Risk factors for NAFLD among patients with CKD have only been investigated in small-scale studies with often inadequate methods. No studies have investigated the impact of fat lipid content measured by MR spectroscopy in patients with type 2-diabetes and CKD stage 3-5. New therapeutic strategies for the diagnosis and management of NAFLD in patients with CKD with diabetes are needed and important challenges in the elucidation of the ethology, pathogenesis and prevalence of NAFLD in CKD patients exist.Thus, this project will bring new knowledge among a group of patients with high morbidity and an increased risk of mortality - a knowledge that may provide new guidelines for prevention and treatment of NAFLD.

Objectives

The primary objective of this project is to study the association between the kidney function and the prevalence of NAFLD and the association with type 2-diabetes.

Furthermore, secondary objectives are to investigate potential associations between NAFLD in type 2-diabetes CKD patients and glucose profiles, metabolomics- and lipidomics profiles, intestinal peptides and the bile acid metabolism.

METHODS

Study design and population

This is a cross-sectional cohort study involving 54 patients with type 2-diabetes with normal kidney function and 54 patients with type 2-diabetes and CKD stage 3-5 (not on dialysis).

The patients will be recruited from the outdoor clinic of either endocrinology or nephrology at Rigshospitalet, Herlev Hospital, Steno Diabetes Center Copenhagen and Gentofte Hospital.

Examinations

The project involves following methods.

Magnetic resonance (MR) spectroscopy Fibroscan and clinical index Blood samples Dual Energy X-ray Absorptiometry scan Continuous Glucose Monitoring Clinical examination

Data and statistical analysis

The null hypothesis is that there is no difference in relative liver lipid signal measured by MR spectroscopy between type 2-diabetic patients with CKD stage 3-5 and patients with type 2-diabetes and normal renal function.

The alternative hypothesis is that there is a difference of 30% in liver lipid signal between type 2-diabetic patients with CKD stage 3-5 and patients with type 2-diabetes and normal renal function. In the literature content in relative liver fat signal in patients with type 2-diabetes and CKD 3-5 is about 60% and in type 2-diabetes patients with normal function it is about 30%. In a two-sided t-test with α=0.05 and power of 80%, a sample size of 98 patients in a parallel design is needed to demonstrate a difference in relative liver fat signal between type 2-diabetes patients with CKD 3 and 5 and type 2 diabetes patients with normal renal function of 30%. A total of 108 patients, including 10 extra patients, are planned to be examined.

After completion of the study and data completion the results are analysed according to primary and secondary endpoints. Results are reported as mean values with confidence interval or median and range. Data are analysed with parametric (normally distributed data) or non-parametric statistics (non-normal distributed data). A 95 % confidence interval is accepted as statistically significant (p < 0.05).

All data will be pseudo anonymised.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosed type 2-diabetes
* eGFR > 60 ml/ min/ 1,73 m2 with absence of proteinuria (N=54) OR eGFR < 60 ml/ min/ 1,73 m2 (N=54)
* Outpatient at the department of endocrinology at either Rigshospitalet, Herlev Hospital, Gentofte Hospital or Steno Diabetes Center Copenhagen OR Outpatient at the department of nephrology at either Rigshospitalet or Herlev Hospital

EXCLUSION CRITERIA

* End stage liver disease as diagnosed by MELD (model for end stage liver disease) criteria OR
* At the waiting list for liver transplantation OR
* Daily alcohol intake above 20 g and 30 g for women and men respectively OR
* Known hepatitis A, B or C or hepatocellular carcinoma or other known liver disease OR
* Dialysis therapy OR
* Pregnancy OR
* Weight > 130 kg OR
* Implanted pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Total number of participants: 108 divided in two Groups:
  * 54 patients with diabetes type 2 and normal kidney function (eGFR >60 and absense of clinical proteinuria)
  * 54 patients with diabetes type 2 and chronic kidney disease stage 3-5
  The patients are recruited from the department of Endocrinology or Nephrology at Rigshospitalet (if necessary, from Herlev Hospital, Gentofte Hospital or Steno Diabetes Center Copenhagen also).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Prevalence of NAFLD and actual estimate of liver signal measured by MR spectroscopy | 1 day
  Liver signal is measured by MR spectroscopy

SECONDARY OUTCOMES:
Prevalence and actual estimate of liver lipid signal measured by MR spectroscopy in relation to bile acids measured in the blood | 2 visits - MR spectroscopy one day, blood samples another day.
  Liver lipid signal measured by MR spectroscopy. Bile acids are measured and analysed from blood samples.
NAFLD, as measured by MR spectroscopy, and its association with metabolomics and lipidomic profiles measured in the blood in relation to impaired renal function | 1 day
  Measured by blood samples.
The prevalence of fibrosis | 1 day
  As determined by fibroscan of the liver.
NAFLD, as measured by MR spectroscopy, and its association with glucose profiles in relation to impaired renal function | 4 days
  Continuous Glucose Monitoring is used.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-Rasmussen, Professor, Principal Investigator — Department of Nephrology, Rishospitalet, University of Copenhagen
Locations (1):
- Department of Nephrology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No